CLINICAL TRIAL: NCT06573359
Title: Turkish Validity and Reliability of the Expanded Rehabilitation Complexity Scale in Patients in the Stroke Palliative Care Unit
Brief Title: Turkish Validity and Reliability of the Expanded Rehabilitation Complexity Scale
Status: Recruiting | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Sedef Ersoy, MD, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: IstanbulPMRTRHSE
Record Dates: First submitted 2024-08-24; First posted 2024-08-27 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: Rehabilitation Complexity Scale; needs assessment
MeSH Terms: conditions — Stroke | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Turkish translation of the scale will be made by a native English speaker and the back translation will be made into English, and the consistency of the original and Turkish translation will be evaluated by a three-person expert committee. The psychometric properties of the scale will be investigated according to the methods used for the validity of the original scale. The validity of the scale was validated by analyzing the correlations between the rcs-e-tr score obtained at admission (both for each partial item and the total score) and other suitability indicators used in Turkey (FIM Motor and Barthel) using Spearman's rank correlation coefficient r (rho). will be evaluated. Additionally, to check the ability of rcs-e-tr to capture case complexity, it will be correlated with other scores usually recorded in our rehabilitation services on admission, using Spearman's rank correlation coefficient r(rho).

SUMMARY:
The RCS is a tool that can assess the need for complex rehabilitation and objectively indicate that a patient may have difficulty functioning well at home or in the community if their medical needs are still high. Among rehabilitation patients, there are still patients with complex needs, even though they have maximized rehabilitation potential. Moreover, RCS can also be useful in highlighting cases of patients becoming seriously ill during the rehabilitation process due to an acute illness such as sepsis, which significantly limits treatment time. This information can be emphasized using RCS data when requesting extended or increased rehabilitation support.

DETAILED DESCRIPTION:
The Rehabilitation Complexity Scale (RCS) is similarly designed to provide a simple measure of the complexity of rehabilitation needs and/or interventions; This can be implemented in a timely manner and takes into account essential care, specialist nursing, therapy and medical interventions. Clauses in the RCS state that care, nursing, therapy and medical input needs are the primary 'causes' of case complexity and (together with length of stay) will ultimately affect a particular individual. Compliance in healthcare processes is a very current issue, with particular emphasis on the individualization of rehabilitation settings. Compliance has been described by WHO as a complex issue with various dimensions and definitions, and these vary between countries. However, most definitions of appropriateness address a set of basic requirements: that care be effective (based on valid evidence); be efficient (cost-effective); and is consistent with the ethical principles and preferences of the individual, society or society concerned. It is thought that RCS will meet these needs.The research population will be 110 patients selected from the patients hospitalized in the palliative unit of Istanbul Physical Therapy and Rehabilitation Hospital.The sample size was determined as 110. MEDCALC program was used in the analysis. Linear regression analysis was performed. Cronbach-alpha was calculated as 97%.Stabil subacute stroke patients will be included in the study. Barthel, FIM, RCS-E tools will be used in the study.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnoses of stroke -

Exclusion Criteria: unstable cardiac and neurovascular disease

-

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients with subacute(2-6 weeks) stroke
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-08-24 (Actual); Primary Completion 2024-12-26 (Estimated); Study Completion 2025-01-07 (Estimated)

PRIMARY OUTCOMES:
Turkish validation and reliability of the Rehabilitation Complexity Scale (RCS-E) | 1 week for test retest interrater and intrarater evaluation. 2 months for the study
  The validity of the scale was validated by analyzing the correlations between the rcs-e-tr score obtained at admission (both for each partial item and the total score) and other suitability indicators used in Turkey (FIM Motor and Barthel) using Spearman's rank correlation coefficient r (rho). Additionally, to check the ability of rcs-e-tr to capture case complexity, it will be correlated with other scores usually recorded in our rehabilitation services on admission, using Spearman's rank correlation coefficient r(rho). Files will be viewed simultaneously and independently in a blinded manner by three researchers to assess the reproducibility of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: sedef ersoy, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Research and Training Hospital, Istanbul, Bahçelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 months